CLINICAL TRIAL: NCT01194076
Title: Wait-list Feasibility Study of One-Week Intensive Cognitive-Behavioral Therapy for Pediatric OCD
Brief Title: Wait-list Study of One-Week Intensive Cognitive-Behavioral Therapy for Pediatric Obsessive-Compulsive Disorder (OCD)
Acronym: 5dayOCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of South Florida (Other); Fordham University (Other)
Responsible Party: Principal Investigator, Stephen Whiteside, PHD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0082590
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Obsessive Compulsive Disorder
Keywords: cognitive behavior therapy; exposure and response prevention; pediatric; obsessive compulsive disorder; child; anxiety; intensive; OCD; CBT
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5day intensive treatment (Experimental)
  Interventions: Behavioral: 5-day intensive treatment

INTERVENTIONS:
Behavioral: 5-day intensive treatment — Exposure Based Cognitive Behavioral Therapy administered in 10 appointments over 5 days with an added focus on training parents to be exposure coaches

SUMMARY:
The purpose of this study is to examine how well intensive cognitive-behavioral therapy (CBT) delivered over 5 days works in reducing Obsessive-Compulsive Disorder (OCD) symptoms in children and adolescents. Treatment will consist of exposure and response prevention with an added focus on teaching parents to be exposure coaches.

DETAILED DESCRIPTION:
Although cognitive-behavioral therapy (CBT) is the most effective intervention for pediatric obsessive-compulsive disorder (OCD), many people do not receive CBT initially due, in part, to the lack of trained providers and geographic barriers (e.g., distance to such providers). Rather, the majority of youth with OCD receive psychiatric medication alone or together with unproven forms of psychotherapy. While some serotonergic medications have demonstrated utility in pediatric OCD, side effects can be common, response rates are modest at best, and symptom remission is rare. Storch et al. have shown that CBT can be delivered effectively in an intensive format over a 3-week time-span; however, even this shortened treatment approach involves considerable time and financial expenditure for those who do not have local access to CBT, including three week's time off from work and the cost of local room and board. Given this, more efficient ways of providing CBT need to be identified and tested to increase the number of people with access to this form of treatment. With this in mind, the proposed feasibility study examines the use of videophone technology to evaluate a 5-day cognitive-behavioral intervention for youth with OCD administered at multiple sites. A total of 30 youth will receive 10 60-75-minute sessions of CBT over 5 days (two sessions a day). Cognitive-behavioral therapy will be based on a demonstrated effective treatment protocol, and adapted for administration over a one-week time-span. We will utilize a month-long waitlist control to estimate treatment efficacy. Comprehensive assessments will be conducted by trained clinicians at relevant time-points (i.e., baseline, post-waitlist, post-treatment, follow-up) to assess symptom severity and impairment. Should supporting data be found, CBT delivered in a 5-day format would have the potential to help many more families who would otherwise remain untreated or inadequately treated.

ELIGIBILITY:
Inclusion Criteria:

* All patients must meet the following inclusion criteria to be eligible for study participation:

  * Principal diagnosis of OCD on the ADIS-IV-P and CY-BOCS Total Score ≥ 16
  * No change in psychotropic medication (if applicable) for at least 8 weeks prior to study entry
  * 7 to 17 years old
  * Availability of at least one parent to accompany the child to all assessment sessions and be present for videophone assessments
  * Have a computer and high-speed internet within their home
  * English speaking.

Exclusion Criteria:

* Patients will be excluded from the study if they meet any of the following criteria:

  * History of and/or current psychosis, autism, bipolar disorder, or current suicidality, oppositional defiant disorder, or eating disorder measured by the ADIS-IV-P and all available clinical information
  * Principal diagnosis other than OCD
  * Current a positive diagnosis in the caregiver of mental retardation, psychosis, or other psychiatric disorders or conditions that would limit their ability to understand CBT (based on clinical interview).
* Participants can be included if they are taking a selective serotonin reuptake inhibitor, SNRI, tricyclic, or antipsychotic provided that no medication changes were made 8 weeks prior to initiation of CBT or during treatment.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Children's Yale Brown Obsessive Compulsive Scale (CYBOCS) | 1 month before tx, pre-tx, post-tx, 3 month follow-up
  The CYBOCS is the gold standard measure of OCD symptoms. The primary outcome is the decrease in CYBOCS scores from pre-tx to post-tx, and post-tx to follow-up, compared to the change from 1 month before tx to pre-tx.

SECONDARY OUTCOMES:
Spence children's anxiety scale | baseline, pre-tx, post-tx, 3 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Whiteside, PhD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - University of South Florida, Tampa, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Fordham University, The Bronx, New York